CLINICAL TRIAL: NCT01011634
Title: A Double Blinded, Placebo-controlled Randomized Control Trial Comparing Intravenous Moderate Sedation and Oral/Sublingual Analgesia/Anxiolysis for First Trimester Surgical Abortions
Brief Title: Trial Comparing Intravenous and Oral Moderate Sedation for First Trimester Surgical Abortions
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: 7% enrollment. Study terminated after a small number of recruited patients
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H10873-28990-01
Record Dates: First submitted 2009-11-09; First posted 2009-11-11 (Estimated); Results first posted 2013-05-16 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Undesired Intrauterine Pregnancy; First Trimester Pregnancy
Keywords: abortion; uterine aspiration; pain control
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Moderate sedation (Active Comparator)
  Interventions: Drug: Intravenous moderate sedation versus oral medication
- Oral medication (Active Comparator)
  Interventions: Drug: Intravenous moderate sedation versus oral medication

INTERVENTIONS:
Drug: Intravenous moderate sedation versus oral medication — Intravenous moderate sedation (fentanyl 100 mcg and midazolam 2 mg) versus oral analgesia/anxiolysis (lorazepam 2 mg sublingual, hydrocodone/acetaminophen 5/500 mg, and ibuprofen 800 mg)

SUMMARY:
In the United States, the majority of first-trimester surgical abortions are performed in outpatient clinics that utilize a wide variety of oral and intravenous regimens for pain control. The specific aim of this study is to evaluate the equivalency of intravenous moderate sedation (fentanyl 100 mcg and midazolam 2 mg) versus oral analgesia/anxiolysis (lorazepam 2 mg sublingual, hydrocodone/acetaminophen 5/500 mg, and ibuprofen 800 mg) for first-trimester surgical abortions. The investigators hypothesize that oral moderate sedation and intravenous moderate sedation will be equivalent in controlling pain as measured by a difference of +/- 10 on a 100-point (range 0-100) visual analog pain scale.

DETAILED DESCRIPTION:
Approximately 50% of pregnancies in the United States are unintended and about 50% of these end in an induced abortion. In 2000, approximately 1.31 million abortions were performed in the United States, approximately 88% of which were less than 12 weeks gestational age. There has been a movement toward performing elective abortions in the ambulatory care setting; however this can provide a dilemma in terms of the procedural anesthesia. In fact, general anesthesia for induced abortions has been associated with an increased incidence of complications and death.5

The paracervical block (PCB) alone has been shown to reduce pain from cervical dilation and tenaculum placement. Slower injection and greater volume have been associated with greater pain control, possibly related to an effect on tissue distension as well as to nerve blockade.6,7,8 However, women's perception of pain continues to be significant with PCB alone.

A majority of high-volume first trimester providers (abortion clinics) offer intravenous moderate sedation. However, many individual practitioners are limited in their ability to provide outpatient moderate sedation, and research has shown mixed results about its efficacy. There continues to be a dilemma in terms of what constitutes optimal anesthesia for first trimester abortions to maximize pain control and minimize side effects and duration of hospital/clinic stay for the patients. A randomized, double blind, placebo controlled trial of intravenous fentanyl (50-100 mcg) with local anesthesia versus placebo and local anesthesia alone in 368 participants found that fentanyl, when compared with placebo, reduced the pain of first trimester abortion by 1.0 point on an 11-point verbal numerical scale. The investigators concluded that this pain reduction was of questionable clinical significance and less than what study participants desired (2.0 points). Another randomized, double blind, placebo controlled study in 100 participants compared local anesthesia alone to local anesthesia with intravenous fentanyl (25mcg) and midazolam (2mg) for first trimester suction curettage. There was no statistically significant difference in pain scores between the groups. However, patients who received intravenous sedation reported increased satisfaction with their abortion procedure.11

There is some evidence of good pain control with oral and sublingual analgesia. Preliminary data from a study performed at the UCSF Mt. Zion Women's Options Clinic between 11/04 and 12/05 (Meckstroth H10873-25519) of 120 women undergoing first trimester abortions who received sublingual lorazepam, ibuprofen, and cervical block revealed that 84.5% of patients reported their pain as acceptable during the procedure with 4.8% considering their pain level unacceptable and 10.7% unsure.

Considering barriers to abortion access, developing an adequate medication regimen that does not require the monitoring and expense of moderate sedation could be very helpful in encouraging more providers to offer abortion. . Given that many patients pay directly for abortions, increasing the cost of services can be prohibitive for many women. Oral medications may also be more appealing to patients seeking sedation but who are fearful of needles. We hope to demonstrate that pain will be adequately controlled with sublingual lorazepam and oral ibuprofen- ideal medications for the clinic setting.

Currently, the standard of care in the SFGH Women's Option Center is moderate sedation with IV fentanyl and midazolam. We will conduct a randomized control trial to evaluate moderate sedation vs. sublingual lorazepam, oral ibuprofen, and hydrocodone/acetaminophen to assess pain control and satisfaction in patients undergoing first trimester abortions. Both groups will receive local cervical block analgesia.

The proposed study is a randomized, double-blind, controlled trial to be conducted at the San Francisco General Hospital (SFGH) Women's Options Center evaluating the equivalency of intravenous moderate sedation (fentanyl 100 mcg plus midazolam 2 mg) vs oral analgesia/anxiolysis (lorazepam 2 mg sublingual, hydrocodone/acetominophen 5/500 mg, and ibuprofen 800 mg) for first trimester surgical abortions.

The study participants will be derived from the SFGH Women's Options Center. On average, the SFGH Women's Options Center performs about 2200 abortions per year, of which 50% are in the first trimester, and intravenous moderate sedation is currently the standard pain control regimen, utilized in nearly 100% of procedures. In the SFGH's sister clinic at Mt. Zion and at Planned Parenthood Golden Gate and its affiliates, various regimes of oral analgesia/anxiolysis are utilized instead. Both are considered standard of care for early abortion both locally and nationally.

ELIGIBILITY:
Inclusion Criteria:

1. Intrauterine pregnancy <12 weeks gestation (as confirmed by ultrasound)
2. Ability to undergo outpatient abortion without an anesthesiologist
3. Age ≥ 16 years old
4. Informed consent prior to participation in study
5. English or Spanish language capacity (or staff or professional translator available for all study procedures)

Exclusion Criteria:

1. Possible ectopic pregnancy
2. Known allergy to study medications or misoprostol
3. Current unstable psychiatric disorder
4. Current alcohol/drug/narcotic/benzodiazepine/barbituate dependence within the previous 2 months
5. Weight < 50 kg

Ages: 16 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2007-05; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pratima Gupta, MD, Principal Investigator — University of California, San Francisco; Karen Meckstroth, MD, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Moderate Sedation | Oral Medication
Started | 9 | 9
Completed | 9 | 8
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderate Sedation | Oral Medication | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Customized [Number; unit: participants] — no baseline measurement as study stopped for low enrollment
  participants
    >= 18 years old | 9 | 9 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Secondary Outcome: Acceptability of Pain, Would They Choose the Same Regimen Again for Another Uterine Aspiration
Time Frame: 30 min after procedure
Population: Study was stopped due to low enrollment (7%). No data analysis performed.
Arm/Group | Moderate Sedation | Oral Medication
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Pain Score Within 5 Mins After Procedure
Time Frame: within 5 mins after procedure
Population: Study was stopped due to low enrollment (7%). No data analysis performed.
Arm/Group | Moderate Sedation | Oral Medication
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Oral Medications | IV Medications
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No